CLINICAL TRIAL: NCT06492720
Title: A Pilot, Open-label, Two-arm, Parallel-group Randomized Trial Study to Evaluate the Efficacy and Safety of NaviFUS™ System Neuromodulating Treatment for Patients With Drug Resistant Epilepsy
Brief Title: A Pilot Study to Evaluate the Efficacy and Safety of NaviFUS™ System Neuromodulating Treatment for Patients With Drug Resistant Epilepsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NaviFUS Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NF-2023-02
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Drug Resistant Epilepsy; Epilepsy; Epilepsy, Temporal Lobe
Keywords: NaviFUS System; Focused Ultrasound; Low-Intensity Focused Ultrasound; LIFU
MeSH Terms: conditions — Drug Resistant Epilepsy; Epilepsy; Epilepsy, Temporal Lobe | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose group FUS treatment (Experimental): FUS treatment will be conducted with following exposure parameters:
  intracranial spatial-peak temporal-average intensity (ISPTA) ceiling level: 2.8 W/cm2, burst length: 3 ms, duration: three consecutive 5-minute FUS exposures with two 5-minute intermission intervals.
  Interventions: Device: Focused ultrasound (FUS) treatment
- High dose group FUS treatment (Experimental): FUS treatment will be conducted with following exposure parameters:
  intracranial spatial-peak temporal-average intensity (ISPTA) ceiling level: 2.8 W/cm2, burst length: 3 ms, duration: three consecutive 10-minute FUS exposures with two 5-minute intermission intervals.
  Interventions: Device: Focused ultrasound (FUS) treatment

INTERVENTIONS:
Device: Focused ultrasound (FUS) treatment — The mechanism of action of FUS neuromodulation involves the activation of voltage-gated ion channels to induce temporary neuromodulation.

SUMMARY:
This will be a prospective, pilot, open-label, two-arm, parallel-group, randomized study to evaluate the efficacy and safety of low-intensity focused ultrasound (LIFU) neuromodulation using NaviFUS System in patients with drug-resistant epilepsy (DRE).

DETAILED DESCRIPTION:
The study aims to demonstrate the efficacy and safety of LIFU neuromodulation in DRE patients, showing its ability to decrease targeted neuronal activity and alleviate epileptic seizures.

Drug-resistant epilepsy (at least 3 anti-seizure medication failed) patients whose epileptogenic foci have been determined by comprehensive presurgical evaluation and meet all eligibility criteria may participate in this study by providing informed consent. Eligible patients will undergo a 8-week baseline observation screening period and will be asked to keep a 8-week seizure diary. This diary will serve as a baseline prior to treatment and will continue to be recorded throughout the treatment and follow-up period.

This study will enroll a maximum of 16 eligible patients. Eligible patients will be randomized into two groups to receive three-consecutive 5-minute twice (low dose group) or three-consecutive 10-minute FUS treatment twice (high dose group) in a week using assigned ultrasound exposure doses generated by the NaviFUS System. Following treatment, there will be a 24-week follow-up period. Patients will be allowed concomitant use of anti-seizure medications (ASMs) throughout the whole study period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged over than and equal to 18 years old.
2. Patients with drug-resistant epilepsy (defined as at least 3 ASM failed) and 1-4 ASM at the time of study entry.
3. Epileptogenic focus (or foci) is determined by comprehensive presurgical evaluation.
4. At least 4 focal-onset seizures with objectively visible or significantly disabling manifestations in the 8-week baseline and at least one seizure per month in the baseline.
5. Willing and able to sign written informed consent and be able to comply with the study protocol during the study period.

Exclusion Criteria:

1. Patients with concurrent active psychiatric or mood disorders that have been assessed to interfere with participation in the study.
2. Presence of pacemaker, implantable cardioverter-defibrillator (ICD), permanent medication pumps, cochlear implants, or deep brain stimulation (DBS).
3. The skull bone area traversed by the sonication pathway is covered by scars, scalp disorders (e.g., eczema), wounds, or atrophy of the scalp.
4. Image documented calcified lesion in the FUS exposure path.
5. Abnormal coagulation profile:

   1. Platelet (PLT) < 100,000/μL.
   2. prothrombin time (PT) > 15 sec.
   3. activated partial thromboplastin time (APTT) > 45 sec.
   4. international normalized ratio (INR) > 1.5.
   5. Patients requiring anticoagulant medications.
6. Pregnant or breast-feeding women.
7. Coexisting medical problems of sufficient severity to limit compliance with the study.
8. Known sensitivity/allergy to Magnetic Resonance Imaging (MRI) contrast agents or any of its components; having metallic implants that are assessed as unsuitable for MRI examination.
9. Use of any recreational drugs or history of drug addiction or known history of substance or alcohol abuse.
10. Patients have received an investigational drug or an investigational device within 4 weeks prior to the study
11. Any other condition that, in the investigator's judgment, might affect study endpoints or might increase the risk to the patients or decrease the chance of obtaining satisfactory data needed to achieve the objectives of the study.
12. Any ASM treatment change during the baseline (screening period).
13. Vagus nerve stimulation (VNS) dosing changes within 2 months before baseline (screening period).
14. Radiofrequency thermocoagulation (RFTC) within 2 months before baseline (screening period).
15. Patient has an IQ < 70, based on the Wechsler Abbreviated Scale of Intelligence (WASI-III or IV).
16. Any other condition that, in the investigator's judgment, patient not applicable to participate this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-08-10 (Estimated)

PRIMARY OUTCOMES:
Changes of seizure frequency after treatment compared to baseline | up to 33 weeks
  The changes in patient's seizure frequency from baseline through the study completion will be assessed based on the seizure diaries.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | up to 33 weeks
  The incidence and severity of AEs associated with LIFU neuromodulation in patients with DRE.
Responder rate (≧50% seizure reduction) | up to 33 weeks
  The changes in responder rate (≧50% seizure reduction) from baseline through the study completion will be assessed based on the seizure diaries.
Change from baseline in number of seizure-free days | up to 33 weeks
  The changes in number of seizure-free days from baseline through the study completion will be assessed based on the seizure diaries.
Change from baseline in subjective seizure strength | up to 33 weeks
  The changes in subjective seizure strength from baseline through the study completion will be assessed based on the seizure diaries.
Quality of Life in Epilepsy (QOLIE-31) | up to 33 weeks
  The QOLIE-31 is a survey of health-related quality of life for adults with epilepsy. There are 31 questions about patient's health and daily activities. The total score is calculated as a weighted mean of the sub-scale scores and the scoring of the QOLIE-31 requires the conversion of raw data to a scale of 0 to 100 for each sub-scale, with higher scores reflecting higher quality of life.
Changes of Beck Anxiety Inventory (BAI) after treatment compared to baseline | up to 33 weeks
  BAI is a 21-question multiple-choice self-report inventory that is used to measure the severity of anxiety. Each answer is scored on a scale value of 0 (not at all) to 3 (severely). Higher total scores indicate more severe anxiety symptoms.
Changes of Beck Depression Inventory (BDI) after treatment compared to baseline | up to 33 weeks
  BDI-II, a 21-question multiple-choice self-report inventory, is a psychological test used to measure the severity of depression. Each answer is rated on a scale of 0 (none at all) to 3 (severe). Higher total scores indicate more severe depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen SG, Tsai CH, Lin CJ, Lee CC, Yu HY, Hsieh TH, Liu HL. Transcranial focused ultrasound pulsation suppresses pentylenetetrazol induced epilepsy in vivo. Brain Stimul. 2020 Jan-Feb;13(1):35-46. doi: 10.1016/j.brs.2019.09.011. Epub 2019 Sep 24. PMID 31575487
- [Background] Chu PC, Yu HY, Lee CC, Fisher R, Liu HL. Pulsed-Focused Ultrasound Provides Long-Term Suppression of Epileptiform Bursts in the Kainic Acid-Induced Epilepsy Rat Model. Neurotherapeutics. 2022 Jul;19(4):1368-1380. doi: 10.1007/s13311-022-01250-7. Epub 2022 May 17. PMID 35581489
- [Background] Lee CC, Chou CC, Hsiao FJ, Chen YH, Lin CF, Chen CJ, Peng SJ, Liu HL, Yu HY. Pilot study of focused ultrasound for drug-resistant epilepsy. Epilepsia. 2022 Jan;63(1):162-175. doi: 10.1111/epi.17105. Epub 2021 Nov 2. PMID 34729772